CLINICAL TRIAL: NCT01255098
Title: A Development Plan of in Vitro Diagnostics of Immuno Magnetic Reduction Assay - A Rapid Etection Kit of Enterobacteraceae in Blood or Blood Culture
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Giueng-Chueng Wang, Laboratory Medicine
Other Study IDs: 98085
Record Dates: First submitted 2010-12-03; First posted 2010-12-07 (Estimated); Last update posted 2010-12-07 (Estimated); Status verified 2010-12

CONDITIONS: Immuno Magnetic Reduction

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Experimental Group
- Control Group

SUMMARY:
This plan is to develop blood culture or to measure diagnostics of Immuno Magnetic Reduction assay in the first stage.

ELIGIBILITY:
Inclusion Criteria:

* emergency cases
* blood culture of positive and negative cases which storage in 4℃ every day

Exclusion Criteria:

* not emergency cases of blood culture

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: emergency cases
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2009-11; Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giueng-Chueng Wang, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University WanFang Hospital, Taipei, Taiwan